CLINICAL TRIAL: NCT03944980
Title: Phase III Clinical Study of PD-1 Monoclonal Antibody-activated Autologous Peripheral Blood T-Lymphocyte (PD1-T) Combined With Docetaxel in the Second-line Treatment of IIIB/IIIC/IV Non-small Cell Lung Cancer
Brief Title: Study of Chemotherapy Combination With Autologous Cell Immunotherapy in the Advanced Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2018-150-01
Record Dates: First submitted 2019-04-28; First posted 2019-05-10 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-04

CONDITIONS: IIIB/IIIC/IV Lung Cancer
Keywords: Effect; Safety
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: CIK (Experimental): Docetaxel & PD1-T cells
  Docetaxel,60mg/m2,intravenous infusion,d1; PD1-T cells, 1x10^10 (10 billion ), intravenous infusion,d14; Q3W.
  Interventions: Drug: Docetaxel; Biological: PD1-T cells
- Arm 2: Control (Active Comparator): Docetaxel
  Docetaxel,60mg/m2,intravenous infusion,d1; Q3W.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Docetaxel injection
Biological: PD1-T cells — PD1-T cells injection
  Other Names: PD-1 monoclonal antibody-activated peripheral blood T-lymphocyte
  Arms: Arm 1: CIK

SUMMARY:
This study evaluates the effect and safty of PD-1 monoclonal antibody-activated autologous peripheral blood T-lymphocyte (PD1-T) combined with docetaxel in the second-line treatment of IIIB/IIIC/IV non-small cell lung cancer. Half of participants receive PD1-T combined with docetaxel, while the other half will receive docetaxel.

ELIGIBILITY:
Inclusion Criteria:

Subjects who must meet all the following criteria should be selected:

1. Agreeing to participate in this study and signing a written informed consent.
2. Male or female,from 18 to 75 years (including 18 and 75 years).
3. The life expectancy is longer than 3 months and can be followed up.
4. Patients with stage IIIB/IIIC/IV NSCLC were confirmed by histological /cytological and imaging examinations. According to RECIST 1.1 standard, there will be at least one measurable lesion.
5. According to RECIST 1.1 standard, the researchers evaluated the pre-test imaging to determine the progression of the disease after at least two cycles of platinum-containing double chemotherapies.
6. ECOG score will be 0 or 1 within 7 days before randomization.
7. Within 14 days before the start of treatment, the results of laboratory test of blood routine, liver, kidney function and hormone levels must be met the following criteria:

   White blood cells: more than 3.0 × 109/L; Platelets: more than 100 × 109/L; Neutrophils: more than 1.5 × 109/L; Hemoglobin: more than 80g/L; Serum glutamate pyruvate transaminase: less than 2.5 folds of the upper normal limit (ULN); Serum glutamic-oxal (o) acetic transaminase: less than 2.5 × ULN; Serum bilirubin: less than 1.25 × ULN; Serum creatinine: less than 1.25 × ULN. Cortisol and thyroid function will be in the normal range.
8. The toxicity and side effects of previous chemotherapy will must be alleviated to grade 1 or below (except hair loss).
9. Female subjects must take effective contraceptive measures throughout the study period; serum or urine pregnancy test results must be negative during screening and the whole study period.
10. Male subjects should take effective contraceptive measures from the beginning of treatment to within 6 months after the end of treatment.

Exclusion Criteria:

Subjects who meet any of the following criteria could not participate in this study:

1. Adenocarcinoma subjects with EGFR sensitive mutation or ALK translocation; molecular detection of EGFR-sensitive mutations or ALK translocations is not required in squamous carcinoma patients.
2. NSCLC that had received docetaxel treatment in the past.
3. Other malignant tumors needed treatment within five years.
4. Allogeneic tissue/organ transplantation.
5. Participating in research drug therapy within 4 weeks before the first administration of the trial.
6. Systemic glucocorticoid therapy or any other form of immunosuppressive therapy (except glucocorticoid preconditioned with docetaxel) is being administered within 3 days before the first administration of the experimental therapy.
7. Received anti-tumor monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy or major surgery within 4 weeks before the first use of the drug; received chest radiotherapy greater than 30 Gy within 6 months before the first use of the drug; and received chest radiotherapy with 30 Gy or less within 1 month before the first use of the drug.
8. Previous treatment with PD-1/PD-L1 antibodies.
9. Over the past two years, patients with active autoimmune diseases requiring systemic treatment, such as the use of corticosteroids, or immunosuppressants. Substitution therapy (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary dysfunction) is not a systemic treatment.
10. Patients with congenital or acquired immunodeficiency (e.g. HIV-infected persons), active hepatitis B (HBV-DNA > 10^3 copies/ml) or hepatitis C (hepatitis C antibody positive), and HCV-RNA higher than the detection limit of the analytical method.
11. Subjects with active central nervous system (CNS) metastases and/or cancerous meningitis.
12. Patients with active infections requiring systemic intravenous therapy.
13. Mental illness or other illnesses, such as uncontrollable heart disease or pulmonary disease, diabetes, etc.
14. Subjects who are known to be allergic to any of the constituents of the drug being studied.
15. Subjects with a recent history of drug abuse (including alcohol) within one year.
16. Compliance is poor and can not cooperate with clinical research.
17. Female subjects who are pregnant or breastfeeding, or who are expected to be pregnant during the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  PFS will be calculated from initiation of treatment until first progression, and patients alive in stable state will be censored at the time of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Xiubao Ren, MD. PhD., Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China